CLINICAL TRIAL: NCT02711956
Title: A Phase 1b/2a Safety and Tolerability Study of ZEN003694 in Combination With Enzalutamide in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of ZEN003694 in Combination With Enzalutamide in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zenith Epigenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEN003694-002
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer (mCRPC); Phase 1b/2a; Prostate Cancer; Pharmacokinetics (PK); ZEN003694; ZEN-3694; Metastatic Castrate-Resistant Prostate Cancer; BET inhibitor (BETi); Bromodomain; Pharmacodynamics (PD); Enzalutamide; XTANDI; MDV3100; Epigenetics
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DE and DC - ZEN003694 in Combination with Enzalutamide (Experimental): Dose Escalation (DE) and Dose Confirmation (DC): ZEN003694 will be administered orally once daily with enzalutamide in 28-day cycles, enrolling mCRPC patients.
  Two patient populations will be enrolled in DE and DC. Cohort A: Patients with prior progression on enzalutamide or apalutamide by PCWG2 criteria who were receiving a stable dose of enzalutamide at the time of study entry. Cohort B: Patients who were enzalutamide-naïve with prior progression on abiraterone by Prostate Cancer Working Group 2 (PCWG2) criteria.
  Interventions: Drug: ZEN003694; Drug: Enzalutamide

INTERVENTIONS:
Drug: ZEN003694
Drug: Enzalutamide
  Other Names: XTANDI; MDV3100

SUMMARY:
This is an open label, non-randomized, Phase 1b/2a, dose escalation and dose confirmation study of ZEN003694 in combination with enzalutamide in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 years
2. Metastatic, castrate resistant, histologically confirmed prostate cancer; surgically castrated or continuous medical castration for ≥ 8 weeks prior to screening
3. Serum testosterone < 50 ng/dL determined within 4 weeks of first administration of study drug
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Adequate laboratory parameters [absolute neutrophil (ANC), platelets, asparate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, creatinine and coagulation parameters] at screening
6. Dose Escalation Cohort DE-A: Prior progression on enzalutamide or apalutamide at any time by PCWG2 criteria and receiving a stable dose of enzalutamide at the start of study treatment.
7. Dose Escalation Cohort DE-B: Enzalutamide-naïve and apalutamide-naïve patients following prior progression on abiraterone by PCWG2 criteria and receiving a stable dose of enzalutamide at the start of study treatment.
8. Dose Confirmation Cohort A (DC-A) only: Currently receiving enzalutamide as most recent systemic therapy for mCRPC and have experienced PSA progression by PCWG2 criteria in the absence of radiographic and/or clinical progression. Patients may or may not have experienced prior progression on abiraterone.
9. Dose Confirmation Cohort B (DC-B) only: Enzalutamide-naïve patients following prior progression on abiraterone by PCWG2 criteria and within 12 weeks of discontinuing abiraterone.

Exclusion Criteria:

1. Any history of brain metastases or prior seizure or conditions predisposing to seizure activity
2. Have previously received an investigational BET inhibitor (including previous participation in this study or Study ZEN003694-001)
3. Have received prior systemic anti-cancer therapy (including abiraterone) or investigational therapy within 2 weeks or five half-lives, whichever is shorter, prior to the first administration of study drug
4. Failure to recover to Grade 1 or lower toxicity related to prior systemic therapy (excluding alopecia and neuropathy) prior to study entry
5. Radiation therapy within 2 weeks of the first administration of study drug
6. Have received prior chemotherapy in the metastatic castration-resistant setting (prior chemotherapy in the hormone-sensitive setting is allowed provided last dose was at least 6 months prior to study entry)
7. Have received prior investigational anti-androgen therapy, including ARN-509
8. Currently receiving medications known to be strong inhibitors of CYP2C8, strong inducers (except enzalutamide) or inhibitors of CYP3A4 and substrates of CYP3A4, CYP2C9 and CYP2C19 with a narrow therapeutic window. Strong inducers, inhibitors and substrates must be discontinued at least 7 days prior to the first administration of study drug.
9. Not a candidate for enzalutamide treatment, in the opinion of the Investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine - New York Presbyterian, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at seven investigational sites in the United States between December 2016 and November 2019
Pre-assignment Details: 75 participants were enrolled and treated in the study.
Groups:
- DE-A - 48 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-A - 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-A - 72 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (72 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-A - 96 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-A - 120 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (120 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-A - 144 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B - 36 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B - 48 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B - 72 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (72 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B 96 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-A 48 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-A 96 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles
- DC-B 48 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles
- DC-B 96 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles
Period: Overall Study
Arm/Group | DE-A - 48 mg ZEN003694 + Enzalutamide | DE-A - 60 mg ZEN003694 + Enzalutamide | DE-A - 72 mg ZEN003694 + Enzalutamide | DE-A - 96 mg ZEN003694 + Enzalutamide | DE-A - 120 mg ZEN003694 + Enzalutamide | DE-A - 144 mg ZEN003694 + Enzalutamide | DE-B - 36 mg ZEN003694 + Enzalutamide | DE-B - 48 mg ZEN003694 + Enzalutamide | DE-B 60 mg ZEN003694 + Enzalutamide | DE-B - 72 mg ZEN003694 + Enzalutamide | DE-B 96 mg ZEN003694 + Enzalutamide | DC-A 48 mg ZEN003694 + Enzalutamide | DC-A 96 mg ZEN003694 + Enzalutamide | DC-B 48 mg ZEN003694 + Enzalutamide | DC-B 96 mg ZEN003694 + Enzalutamide
Started | 2 | 2 | 3 | 5 | 4 | 3 | 4 | 4 | 4 | 3 | 1 | 9 | 17 | 6 | 8
Completed | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not Completed | 2 | 2 | 2 | 3 | 4 | 2 | 4 | 2 | 4 | 3 | 1 | 9 | 16 | 5 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 1
Not completed — Clinical progression | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 4 | 1 | 1
Not completed — Radiographic progression | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 3 | 0 | 1
Not completed — PSA progression with clinical progression | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — PSA progression with radiographic progression | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All treated safety population consisted of all treated participants.
Groups:
- DE-B - 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE-B - 96 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-A - 48 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-A - 96 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-B - 48 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DC-B - 96 mg ZEN003694 + Enzalutamide: Dose Confirmation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | DE-A - 48 mg ZEN003694 + Enzalutamide | DE-A - 60 mg ZEN003694 + Enzalutamide | DE-A - 72 mg ZEN003694 + Enzalutamide | DE-A - 96 mg ZEN003694 + Enzalutamide | DE-A - 120 mg ZEN003694 + Enzalutamide | DE-A - 144 mg ZEN003694 + Enzalutamide | DE-B - 36 mg ZEN003694 + Enzalutamide | DE-B - 48 mg ZEN003694 + Enzalutamide | DE-B - 60 mg ZEN003694 + Enzalutamide | DE-B - 72 mg ZEN003694 + Enzalutamide | DE-B - 96 mg ZEN003694 + Enzalutamide | DC-A - 48 mg ZEN003694 + Enzalutamide | DC-A - 96 mg ZEN003694 + Enzalutamide | DC-B - 48 mg ZEN003694 + Enzalutamide | DC-B - 96 mg ZEN003694 + Enzalutamide | Total
Number analyzed (Participants) | 2 | 2 | 3 | 5 | 4 | 3 | 4 | 4 | 4 | 3 | 1 | 9 | 17 | 6 | 8 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (0.71) | 63.0 (1.41) | 69.0 (18.03) | 62.6 (10.26) | 66.5 (5.80) | 73.0 (3.61) | 73.8 (3.50) | 65.5 (11.33) | 75.0 (13.49) | 67.0 (12.49) | 62 | 67.9 (9.20) | 71.2 (7.59) | 68.2 (6.71) | 71.3 (7.98) | 69.2 (8.68)
Age, Continuous [Median (Full Range); unit: years] | 69.5 [69 to 70] | 63 [62 to 64] | 74 [49 to 84] | 63 [47 to 74] | 67.5 [59 to 72] | 72 [70 to 77] | 73.5 [70 to 78] | 63.5 [54 to 81] | 74.5 [62 to 89] | 71 [53 to 77] | 62 | 66 [52 to 82] | 70 [59 to 83] | 67 [61 to 77] | 72 [57 to 84] | 70 [47 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 3 | 5 | 4 | 3 | 4 | 4 | 4 | 3 | 1 | 9 | 17 | 6 | 8 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 7
  Not Hispanic or Latino | 1 | 2 | 3 | 4 | 4 | 3 | 4 | 4 | 4 | 2 | 1 | 8 | 16 | 6 | 6 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
  White | 1 | 2 | 3 | 4 | 4 | 3 | 4 | 3 | 4 | 2 | 1 | 7 | 11 | 6 | 8 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 4
Mean Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI not available for one participant in DC-A 48 mg
  kg/m^2
    number analyzed (Participants) | 2 | 2 | 3 | 5 | 4 | 3 | 4 | 4 | 4 | 3 | 1 | 8 | 17 | 6 | 8 | 74
    (all) | 25.26 (1.854) | 38.54 (0.882) | 27.18 (5.505) | 29.01 (5.201) | 33.99 (6.138) | 32.58 (6.447) | 25.91 (1.557) | 29.74 (6.805) | 30.25 (6.699) | 27.54 (0.825) | 34.87 | 28.1 (3.763) | 26.05 (4.183) | 28.13 (2.523) | 28.34 (3.670) | 28.54 (4.895)
Median Body Mass Index [Median (Full Range); unit: kg/m^2] — Population: BMI not available for one participant in DC-A 48 mg
  kg/m^2
    number analyzed (Participants) | 2 | 2 | 3 | 5 | 4 | 3 | 4 | 4 | 4 | 3 | 1 | 8 | 17 | 6 | 8 | 74
    (all) | 25.26 [24.0 to 26.6] | 38.54 [37.9 to 39.2] | 27.8 [21.4 to 32.3] | 29.24 [22.3 to 36.7] | 32.83 [28.0 to 42.3] | 29.49 [28.2 to 40.0] | 25.98 [24.2 to 27.5] | 29.02 [22.3 to 38.6] | 29.62 [22.8 to 38.9] | 27.53 [26.7 to 28.4] | 34.87 | 27.09 [24.2 to 36.4] | 25.81 [21.2 to 39.2] | 27.66 [25.2 to 32.5] | 29.38 [23.8 to 32.7] | 27.69 [21.2 to 42.3]
Mean PSA [Mean (Standard Deviation); unit: ng/mL] | 37.295 (17.9534) | 96.855 (132.7452) | 10.383 (7.8450) | 8.996 (7.0365) | 90.718 (87.1840) | 6.280 (4.7483) | 149.423 (157.4893) | 34.766 (10.52727) | 53.404 (21.9723) | 24.433 (5.2254) | 12.720 | 38.358 (41.2016) | 167.043 (274.6941) | 112.449 (185.2442) | 88.141 (78.4200) | 84.364 (156.2876)
Median PSA [Median (Full Range); unit: ng/mL] | 37.295 [24.6 to 49.99] | 96.855 [2.99 to 190.72] | 8.090 [3.94 to 19.12] | 10.449 [1.12 to 18.77] | 90.850 [6.21 to 174.96] | 5.500 [1.97 to 11.37] | 130.866 [5.42 to 330.54] | 29.881 [28.70 to 50.60] | 53.697 [30.58 to 75.65] | 23.722 [19.60 to 29.98] | 12.720 | 25.600 [0.09 to 116.44] | 29.750 [1.18 to 1079.06] | 52.043 [1.16 to 486.60] | 87.518 [1.48 to 184.24] | 28.700 [0.09 to 1079.06]
ECOG performance status [Count of Participants; unit: Participants] — Classified on a 6-point (0 to 5) rating scale.
  0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5 - Dead
  Participants
    0 | 1 | 1 | 2 | 4 | 3 | 3 | 1 | 3 | 1 | 1 | 1 | 6 | 10 | 4 | 4 | 45
    1 | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 3 | 2 | 0 | 3 | 7 | 2 | 4 | 30

OUTCOME MEASURES:

1. Primary Outcome: For Dose Escalation: Incidence of Dose-limiting Toxicities (DLT) to Determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of ZEN003694 in Combination With Enzalutamide.
Description: Determination of DLT was made during the first 28 days of treatment in the dose escalation phase. A DLT is defined as a clinically significant AE or laboratory abnormality that is considered possibly, probably, or definitely related to study drug. The MTD reflects the highest dose of ZEN003694 in combination with enzalutamide that did not cause a DLT in more than 1 of 6 patients. The RP2D is the recommended dose of ZEN003694 in combination with enzalutamide as determined in the dose confirmation phase of the study.
Time Frame: Cycle 1 (Day 1 thru Day 28)
Population: Participants in dose escalation
Measure: Count of Participants; unit: Participants
Groups:
- DE A+B - 36 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 48 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A+B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 72 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (72 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 96 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 120 mg ZEN003694 + Enzalutamide: Dose Escalation Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (120 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B - 144 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE A+B - 36 mg ZEN003694 + Enzalutamide | DE A+B - 48 mg ZEN003694 + Enzalutamide | DE A+B - 60 mg ZEN003694 + Enzalutamide | DE A+B - 72 mg ZEN003694 + Enzalutamide | DE A+B - 96 mg ZEN003694 + Enzalutamide | DE A+B - 120 mg ZEN003694 + Enzalutamide | DE A+B - 144 mg ZEN003694 + Enzalutamide
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: For Dose Escalation and Dose Confirmation: Incidence of Treatment-emergent Adverse Events (TEAE) and Treatment-related Serious Adverse Events (SAE)
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity of AEs was graded based on the National Cancer Institute's Common Terminology for Adverse Events (V4.03). A serious adverse event (SAE) was any AE that was: fatal; life-threatening; required in-patient hospitalization or prolonged an existing hospitalization; disabling or incapacitating; a congenital anomaly or birth defect; or any other important medical event.
Time Frame: Cycle 1 Day 1 to 30 days post last dose
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- DE - 36 mg ZEN003694 + Enzalutamide: Dose Escalation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC - 48 mg ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE - 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE - 72 mg ZEN003694 + Enzalutamide: Dose Escalation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (72 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC - 96 mg ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE - 120 mg ZEN003694 + Enzalutamide: Dose Escalation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (120 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE - 144 mg ZEN003694 + Enzalutamide: Dose Escalation - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE - 36 mg ZEN003694 + Enzalutamide | DE/DC - 48 mg ZEN003694 + Enzalutamide | DE - 60 mg ZEN003694 + Enzalutamide | DE - 72 mg ZEN003694 + Enzalutamide | DE/DC - 96 mg ZEN003694 + Enzalutamide | DE - 120 mg ZEN003694 + Enzalutamide | DE - 144 mg ZEN003694 + Enzalutamide
Number analyzed (Participants) | 4 | 21 | 6 | 6 | 31 | 4 | 3
Participants
  Blood creatinine increased | 0 | 0 | 2 | 0 | 3 | 0 | 0
  Constipation | 0 | 1 | 0 | 0 | 3 | 0 | 0
  Decreased appetite | 0 | 2 | 2 | 1 | 10 | 3 | 2
  Diarrhea | 0 | 0 | 0 | 1 | 5 | 0 | 0
  Dizziness | 0 | 0 | 0 | 1 | 3 | 0 | 0
  Dysgeusia | 0 | 2 | 0 | 0 | 10 | 1 | 3
  Dyspepsia | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Fatigue | 1 | 8 | 1 | 2 | 13 | 3 | 1
  Nasal congestion | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Nausea | 0 | 7 | 2 | 3 | 17 | 3 | 2
  Photopsia | 0 | 1 | 0 | 0 | 3 | 0 | 0
  Photosensitivity | 0 | 2 | 0 | 0 | 3 | 0 | 0
  Rash | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Rash maculopapular | 0 | 3 | 0 | 0 | 1 | 0 | 1
  Taste disorder | 0 | 0 | 1 | 1 | 3 | 0 | 0
  Thrombocytopenia | 0 | 1 | 1 | 2 | 6 | 0 | 1
  Vision blurred | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Visual symptoms | 3 | 12 | 4 | 6 | 17 | 4 | 2
  Vomiting | 0 | 1 | 0 | 0 | 3 | 1 | 0
  Weight loss and abnormal weight loss | 1 | 0 | 0 | 1 | 3 | 1 | 2

3. Secondary Outcome: Evaluate Prostate-specific Antigen (PSA) Response Rate by PCWG2 Criteria
Description: The PSA response rate will be evaluated using PCWG2 criteria and defined as the proportion of patients with a PSA decline of at least 50%. Any change from baseline is confirmed by a second measurement at least 3 weeks later. PSA Response Rate will be evaluated using PCWG2 criteria and defined as following: Percentage change from baseline in PSA to 12 weeks post ZEN003694 dose. Only evaluate for patients with at least 12 weeks of treatment, the PSA assessment at 12 weeks (84 days +/-3 days) will be used; Maximum percent decrease in PSA from baseline that occurs at any point after treatment. Evaluable for all patients with post-baseline PSA. Arms will be combined to analyze efficacy in Cohort A and Cohort B.
Time Frame: Screening up to 35 months
Population: Arms were combined to analyze efficacy based on Cohorts defined by protocol. Cohort A is defined as patients with prior progression on enzalutamide or apalutamide by PCWG2 criteria. Cohort B is defined as patients who were enzalutamide-naïve with prior progression on abiraterone by PCWG2 criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DE/DC-A ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort A - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 -144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC-B ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 - 96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE/DC-A ZEN003694 + Enzalutamide | DE/DC-B ZEN003694 + Enzalutamide
Number analyzed (Participants) | 45 | 30
percentage of participants | 4.4 [0.5 to 15.1] | 23.3 [9.9 to 42.3]

4. Secondary Outcome: Evaluate Radiographic Response Rate (Overall Response Rate) by PCWG2 Criteria
Description: Tumor response will be evaluated using the PCWG2 criteria. Patients with measurable disease will be evaluated for clinical benefit as determined by tumor response using RECIST v1.1. Patients with non-measurable bone disease will be evaluated for progression based on the presence of any new lesions by bone scans. Radiographic tumor evaluation will be performed at screening and every 3 cycles or more frequently as determined by the investigator. Using the tumor response that is determined by the investigator, best overall response will be determined using RECIST v1.1. Best overall response is defined as the best response recorded from the start of treatment until disease progression or study exit. Arms will be combined to analyze efficacy in Cohort A and Cohort B.
Time Frame: Screening up to 35 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DE/DC A ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort A - Enzalutamide/Apalutamide Progressors - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg - 144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC B ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort B - Abiraterone Progressors - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg - 144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE/DC A ZEN003694 + Enzalutamide | DE/DC B ZEN003694 + Enzalutamide
Number analyzed (Participants) | 39 | 26
percentage of participants | 2.6 [0.1 to 13.5] | 3.8 [0.1 to 19.6]

5. Secondary Outcome: Evaluate Overall Median Progression-free Survival by PCWG2 Criteria
Description: Overall progression free survival (PFS) is determined using the PCWG2 criteria. Overall PFS is measured from screening until the time that disease progression (radiographic progressive disease or clinical deterioration) or death is documented, whichever occurs first. Arms will be combined to analyze efficacy in Cohort A and Cohort B.
Time Frame: Screening up to 35 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DE/DC B ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort B -Abiraterone Progressors - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg - 144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE/DC A ZEN003694 + Enzalutamide | DE/DC B ZEN003694 + Enzalutamide
Number analyzed (Participants) | 45 | 30
months | 4.7 [3.5 to 9.0] | 6.2 [4.6 to 7.9]

6. Secondary Outcome: Evaluate Median Radiographic Progression-Free Survival by PCWG2 Criteria
Description: Radiographic progression-free survival (rPFS) is determined using the PCWG2 criteria to assess both soft-tissue and bone assessments. The rPFS is measured from screening until the time the first radiographic scan shows disease progression, or until the time of death, whichever occurs first. If radiographic disease progression is identified at the first on-treatment radiographic assessment at Cycle 3 Day 1 (8 weeks), radiographic progression must be confirmed by a second assessment 6 or more weeks later. Patients who do not progress radiographically or did not die prior to study exit are censored on the date of their last dose of ZEN003694. Arms will be combined to analyze efficacy in Cohort A and Cohort B.
Time Frame: Screening up to 35 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DE/DC A ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort A - Enzalutamide/Apalutamide Progressors - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg -144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC B ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohort B - Abiraterone Progressors - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg -144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE/DC A ZEN003694 + Enzalutamide | DE/DC B ZEN003694 + Enzalutamide
Number analyzed (Participants) | 45 | 30
months | 10.2 [4.8 to 13.1] | 8.8 [6.1 to 11.5]

7. Secondary Outcome: Measure the Pharmacokinetic (PK) Parameter: AUC(0-24h) of ZEN003694 and ZEN003791 (Active Metabolite) Administered in Combination With Enzalutamide.
Description: AUC(0-24h) is defined as the area under the curve (plasma concentration of drug over a 24-hour time period).
Time Frame: Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose
Population: All Evaluable Participants
Measure: Geometric Mean (Standard Error); unit: ng*h/mL
Groups:
- DE A+B 36 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (36 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC A+B 48 mg ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohorts A+B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 60 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 72 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (72 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE/DC A+B 96 mg ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (96 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 120 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (120 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 144 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A +B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE A+B 36 mg ZEN003694 + Enzalutamide | DE/DC A+B 48 mg ZEN003694 + Enzalutamide | DE A+B 60 mg ZEN003694 + Enzalutamide | DE A+B 72 mg ZEN003694 + Enzalutamide | DE/DC A+B 96 mg ZEN003694 + Enzalutamide | DE A+B 120 mg ZEN003694 + Enzalutamide | DE A+B 144 mg ZEN003694 + Enzalutamide
Number analyzed (Participants) | 4 | 21 | 6 | 6 | 31 | 4 | 3
ng*h/mL
  ZEN003694 AUC(0-24h) Study Day 1 | 1001 (494) | 985 (374) | 2243 (848) | 1966 (1067) | 2424 (1450) | 2153 (1529) | 2119 (1547)
  ZEN003694 AUC(0-24h) Study Day 15; C24 (24h) inputed with Day 15 C0 (pre-dose) for AUC calculations | 867 (651) | 1046 (512) | 1487 (871) | 1453 (967) | 2138 (946) | 2109 (578) | 1641 (704)
  ZEN003791 AUC(0-24h) Study Day 1 | 1335 (659) | 1874 (635) | 3344 (1101) | 3277 (1708) | 4090 (1562) | 3712 (2660) | 3815 (2774)
  ZEN003791 AUC(0-24h) Study Day 15; C24 (24h) imputed with Day 15 C0 (pre-dose) for AUC calculations. | 1234 (606) | 2216 (1187) | 2979 (1583) | 2586 (1265) | 4478 (2449) | 5275 (2369) | 3155 (1858)

8. Secondary Outcome: Measure the Pharmacokinetic (PK) Parameter: Cmax of ZEN003694 and ZEN003791 (Active Metabolite) Administered in Combination With Enzalutamide
Description: Cmax is defined as the maximum or peak plasma concentration of drug.
Time Frame: as for outcome 7
Population: All Evaluable Participants
Measure: Geometric Mean (Standard Error); unit: ng/mL
Groups:
- DE/DC A+B 48 mg ZEN003694 + Enzalutamide: Dose Escalation + Dose Confirmation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (48 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 60 mg ZEN003694 + Enzalutamide PO QD: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (60 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 120 mg ZEN003694 + Enzalutamide PO QD: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (120 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
- DE A+B 144 mg ZEN003694 + Enzalutamide: Dose Escalation - Cohorts A + B - Enzalutamide (160 mg) PO QD 14 days lead-in followed by the combination of ZEN003694 (144 mg) PO QD and enzalutamide (160 mg) PO QD in 28-day cycles.
Arm/Group | DE A+B - 36 mg ZEN003694 + Enzalutamide | DE/DC A+B 48 mg ZEN003694 + Enzalutamide | DE A+B 60 mg ZEN003694 + Enzalutamide PO QD | DE A+B 72 mg ZEN003694 + Enzalutamide | DE/DC A+B 96 mg ZEN003694 + Enzalutamide | DE A+B 120 mg ZEN003694 + Enzalutamide PO QD | DE A+B 144 mg ZEN003694 + Enzalutamide
Number analyzed (Participants) | 4 | 21 | 6 | 6 | 31 | 4 | 3
ng/mL
  ZEN003694 Cmax Study Day 1 | 181 (83) | 216 (103) | 290 (102) | 452 (279) | 492 (277) | 425 (306) | 494 (424)
  ZEN003694 Cmax Study Day 15 | 184 (128) | 236 (119) | 289 (204) | 392 (278) | 484 (189) | 458 (305) | 457 (330)
  ZEN003791 Cmax Study Day 1 | 125 (83) | 184 (62) | 244 (79) | 306 (196) | 374 (143) | 342 (202) | 417 (362)
  ZEN003791 Cmax Study Day 15 | 129 (72) | 220 (101) | 259 (176) | 319 (208) | 477 (194) | 552 (332) | 432 (362)

ADVERSE EVENTS:
Time Frame: For an event to be recorded as an AE, the onset must occur during or after the patient's first exposure to study drug and no later than 30 days after the last study drug dose. There is no limit on reporting SAEs considered reasonably related to ZEN003694.
Description: Adverse events were collected in all participants
Arm/Group | DE A+B 36 mg ZEN003694 + Enzalutamide | DE/DC A+B 48 mg ZEN003694 + Enzalutamide | DE A+B 60 mg ZEN003694 + Enzalutamide | DE A+B 72 mg ZEN003694 + Enzalutamide | DE/DC A+B 96 mg ZEN003694 + Enzalutamide | DE A+B 120 mg ZEN003694 + Enzalutamide | DE A+B 144 mg ZEN003694 + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/21 | 0/6 | 0/6 | 0/31 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 3/21 | 1/6 | 2/6 | 6/31 | 1/4 | 3/3
Other Adverse Events (participants affected / at risk) | 3/4 | 19/21 | 5/6 | 6/6 | 31/31 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE A+B 36 mg ZEN003694 + Enzalutamide (N=4) | DE/DC A+B 48 mg ZEN003694 + Enzalutamide (N=21) | DE A+B 60 mg ZEN003694 + Enzalutamide (N=6) | DE A+B 72 mg ZEN003694 + Enzalutamide (N=6) | DE/DC A+B 96 mg ZEN003694 + Enzalutamide (N=31) | DE A+B 120 mg ZEN003694 + Enzalutamide (N=4) | DE A+B 144 mg ZEN003694 + Enzalutamide (N=3)
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leptospirosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE A+B 36 mg ZEN003694 + Enzalutamide (N=4) | DE/DC A+B 48 mg ZEN003694 + Enzalutamide (N=21) | DE A+B 60 mg ZEN003694 + Enzalutamide (N=6) | DE A+B 72 mg ZEN003694 + Enzalutamide (N=6) | DE/DC A+B 96 mg ZEN003694 + Enzalutamide (N=31) | DE A+B 120 mg ZEN003694 + Enzalutamide (N=4) | DE A+B 144 mg ZEN003694 + Enzalutamide (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 6 | 0 | 1
Visual impairment (Eye disorders) | 3 | 12 | 4 | 6 | 18 | 4 | 2
Photosensitivity reaction (Eye disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 7 | 2 | 3 | 16 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Fatigue (General disorders) | 1 | 9 | 1 | 2 | 13 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 10 | 3 | 2
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 3 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 10 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02711956/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT02711956/SAP_001.pdf